CLINICAL TRIAL: NCT01316133
Title: A Multicenter, Non-comparative, Open-labeled, Prospective Study to Evaluate the Efficacy and Safety of Tacrolimus (Prograf®) With Steroid in Korean Lupus Nephritis Patients Who Are Non-responders to Steroid Monotherapy
Brief Title: A Study to Evaluate the Efficacy and Safety of Tacrolimus With Steroid in Korean Lupus Nephritis Patients
Acronym: APPLE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to poor patient recruitment.
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRGLN-10-01-KOR
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Lupus Nephritis
Keywords: Tacrolimus; Prograf; FK506; Proteinuria; Calcineurin inhibitor
MeSH Terms: conditions — Lupus Nephritis; Proteinuria | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus group (Experimental): Oral
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: Prograf; FK506

SUMMARY:
This study is to evaluate efficacy and safety of tacrolimus with steroid by observing remission rate at 24 weeks in lupus nephritis patients who are non-responders to steroid monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who satisfy more than 4 criteria for diagnosis of systemic lupus erythematosus (ARA criteria, 1982)
* Patients who fall under WHO class III-IV lupus nephritis on renal biopsy
* Patients with refractory lupus nephritis
* Proteinuria ≥ 0.5 g/day
* Patients who took steroid ≥ 20 mg/day over one month prior to the study
* Patients who failed a first-line therapy (non-responders to steroid monotherapy)

Exclusion Criteria:

* Patients who are allergic or resistant to macrolide antibiotics or tacrolimus
* Patients who received tacrolimus in the past (excluding drugs for external use)
* Patients who used other immunosuppressants within 4 weeks before initiation of the study
* Patients who have been receiving systematic chemotherapy since before enrollment (local chemotherapy is allowed.)
* Patients with malignant tumor which developed within the recent 5 years or history of malignant tumor
* Patients who have severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorders which may influence absorption of tacrolimus
* Patients with S-Cr ≥ 200 µ㏖/L or ≥ 2.3 mg/dL
* Patients with liver function levels of more than twice the upper limit of normal or acute active hepatitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-04-19 (Actual); Primary Completion 2016-04-08 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Remission rate | 24 weeks
  Percentage of the patients who shows complete remission or partial remission

SECONDARY OUTCOMES:
Complete remission rate | 24 weeks
Change from baseline in urine protein to creatinine ratio | Baseline, 4 weeks, 12 weeks and 24 weeks
Change from baseline in serum creatinine | Baseline, 4 weeks, 12 weeks and 24 weeks
Safety assessed by the incidence of adverse events, abnormal findings of laboratory tests and vital signs | for 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- South Korea (7):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Seoul

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=209